CLINICAL TRIAL: NCT04781244
Title: Cost-effectiveness of EndWarts® FREEZE for Wart Treatment: A Randomized, Controlled, Investigator-Blinded, Comparative Study
Brief Title: Cost-effectiveness of EndWarts® FREEZE - an Alternative Home Cryotherapy Device for Wart Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EndWart
Record Dates: First submitted 2021-02-25; First posted 2021-03-04 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Cryotherapy Effect; Warts
Keywords: cryotherapy effect; warts; treatment; EndWarts FREEZE
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EndWarts® FREEZE in Soft keratin (Active Comparator): EndWarts® FREEZE were treated to 11 patients with wart at soft keratin
  Interventions: Device: EndWarts® FREEZE
- EndWarts® FREEZE in Hard keratin (Active Comparator): EndWarts® FREEZE were treated to 11 patients with wart at hard keratin
  Interventions: Device: EndWarts® FREEZE
- Liquid nitrogen in Soft keratin (Active Comparator): Liquid nitrogen were treated to 11 patients with wart at soft keratin
  Interventions: Device: Liquid nitrogen
- Liquid nitrogen in Hard keratin (Active Comparator): Liquid nitrogen were treated to 11 patients with wart at hard keratin
  Interventions: Device: Liquid nitrogen

INTERVENTIONS:
Device: EndWarts® FREEZE — EndWarts® FREEZE is an alternative home cryotherapy device. Patients don't have to go to the hospital to receive treatment for their wart.
  Arms: EndWarts® FREEZE in Hard keratin; EndWarts® FREEZE in Soft keratin
Device: Liquid nitrogen — Liquid nitrogen is a conventional cryotherapy treatment for cutaneous wart performed by physician at the hospital.
  Other Names: conventional cryotherapy
  Arms: Liquid nitrogen in Hard keratin; Liquid nitrogen in Soft keratin

SUMMARY:
This study aimed to study cost-effectiveness of EndWarts® FREEZE for wart treatment, compared to conventional liquid nitrogen cryotherapy

DETAILED DESCRIPTION:
Cutaneous warts, caused by Human papilloma virus (HPV), are common skin disease. The prevalence reported in primary school children are 2-20%, and even higher in adults. Non-intact skin are prone to the infection, with all parts of the body can be affected. Even warts are not malignant, they can cause lack of confidence or affected patients' quality of life.

Nowadays there are many treatment methods for warts, such as topical application with salicylic acid and electrical cauterization. Cryotherapy with liquid nitrogen has been the therapy of choice due to its clinical effectiveness, which reported for 6-65%. Treatment mechanism in cryotherapy relies on in-depth freezing of infected keratocyte.

EndWarts® FREEZE is alternative home treatment cryotherapy device containing nitrous oxide. Recent clinical study found that it delivers significant result with good tolerability, and is user friendly. As for our knowledge, no study has been reported about cost-effectiveness of this device, so this study was designed to demonstrate the efficacy of this product in cutaneous warts.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plantar or common wart at Department of Dermatology, Siriraj hospital

Exclusion Criteria:

* Patient with more than 5 warts or wart more than 1 cm in diameter
* Wart at face, genitalia, scalp, joint
* Pregnancy or breastfeeding patient
* Wart with wound/irritation or local infection
* Diabetes mellitus patients or patients with coagulopathies or cryoglobulinemia
* Immunocompromised host or on immunosuppressive drug
* Received any treatment in previous 3 months before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness of EndWarts® FREEZE | 12 weeks
  Evaluate cost-effectiveness of EndWarts® FREEZE for wart treatment compared with conventional liquid nitrogen therapy. Transportation fee to the hospital, medical and doctor fee are recorded to sum up the costs of treatment at every visit. Every patient is also required to have his/her wart examined by the same physician at each visit with the use of dermoscope to evaluate the result of wart treatment (worse, the same, partial response, complete response). Moreover, wart size is measured for its diameter and height, then photographed at each visit to recorded the change after treatment. Cure rates will be shown according to type of intervention received, with the use of chi-square test.

SECONDARY OUTCOMES:
Compared Dermatology quality of life index before and after treatment | 12 weeks
  Compared patient's Dermatology quality of life index (DLQI) between treatment of EndWarts® FREEZE and liquid nitrogen. DLQI is recorded before the treatment start and after 12-week treatment (or before 12 week if the patient's wart is cured completely). Change in DLQI will be shown with descriptive statistics.

OTHER OUTCOMES:
Patient satisfaction of EndWarts® FREEZE | 12 weeks
  Compared patient satisfaction after treatment of EndWarts® FREEZE. Patient who received EndWarts® FREEZE treatment is required to answer the questionnaire after 12-week treatment (or before 12 week if the patient's wart is cured completely). The questionnaire included questions about the opinion of the product, such as effectiveness for wart treatment, portability, user-friendly, safety, and overall satisfaction. Score from each aspect of satisfaction will be calculated with descriptive statistics.
Compared side effect after treatment | 12 weeks
  Compared side effect after treatment with EndWarts® FREEZE and liquid nitrogen. Every patient is required to record his/her side effects after each treatment, such as tingling sensation, burn or scar, hypo/hyperpigmentation, pain, pickling feeling, and report them to the physician at the next follow-up visit (Week 4, week 8, week 12). Number of patients with each side effect are recorded and described with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Charussri Leeyaphan, Assoc. Prof., Principal Investigator — Department of Dermatology Faculty of Medicine, Siriraj Hospital Mahidol University
Locations (1):
- Department of Dermatology, Siriraj Hospital Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Walczuk I, Eertmans F, Rossel B, Cegielska A, Stockfleth E, Antunes A, Adriaens E. Efficacy and Safety of Three Cryotherapy Devices for Wart Treatment: A Randomized, Controlled, Investigator-Blinded, Comparative Study. Dermatol Ther (Heidelb). 2018 Jun;8(2):203-216. doi: 10.1007/s13555-017-0210-5. Epub 2017 Dec 6. PMID 29214505
- [Result] Ghadgepatil SS, Gupta S, Sharma YK. Clinicoepidemiological Study of Different Types of Warts. Dermatol Res Pract. 2016;2016:7989817. doi: 10.1155/2016/7989817. Epub 2016 Mar 7. PMID 27047542
- [Result] Lipke MM. An armamentarium of wart treatments. Clin Med Res. 2006 Dec;4(4):273-93. doi: 10.3121/cmr.4.4.273. PMID 17210977
- [Result] Sterling JC, Gibbs S, Haque Hussain SS, Mohd Mustapa MF, Handfield-Jones SE. British Association of Dermatologists' guidelines for the management of cutaneous warts 2014. Br J Dermatol. 2014 Oct;171(4):696-712. doi: 10.1111/bjd.13310. Epub 2014 Oct 1. No abstract available. PMID 25273231
- [Result] Bruggink SC, Gussekloo J, Berger MY, Zaaijer K, Assendelft WJ, de Waal MW, Bavinck JN, Koes BW, Eekhof JA. Cryotherapy with liquid nitrogen versus topical salicylic acid application for cutaneous warts in primary care: randomized controlled trial. CMAJ. 2010 Oct 19;182(15):1624-30. doi: 10.1503/cmaj.092194. Epub 2010 Sep 13. PMID 20837684